CLINICAL TRIAL: NCT04413032
Title: DreaMS - Development of Digital Biomarkers in Multiple Sclerosis - Feasibility Study
Brief Title: DreaMS - Digital Biomarkers for Multiple Sclerosis
Acronym: DreaMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Research Center for Clinical Neuroimmunology and Neuroscience Basel (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: DreaMS_2020F
Record Dates: First submitted 2020-05-12; First posted 2020-06-02 (Actual); Last update posted 2021-03-02 (Actual); Status verified 2021-03

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Intervention Model Description: A group of patients with Multiple Sclerosis and a group of healthy volunteers will use the dreaMS App over the period of 6 weeks.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with MS (Experimental): 30 Patients with MS will use the DreaMS App over a study duration of 6 weeks.
  Interventions: Device: DreaMS
- Healthy Volunteers (Experimental): 30 Healthy Volunteers will use the DreaMS App over a study duration of 6 weeks.
  Interventions: Device: DreaMS

INTERVENTIONS:
Device: DreaMS — The dreaMS App is a data communication platform collecting data from the patients' mobile devices (smartphone and wearables). We analyze app-based tests, surveys and sensor data.

SUMMARY:
The Investigators have developed the dreaMS App, a data communication platform collecting data from the patients' mobile devices (smartphone and wearables). Through the use of app-based tests, surveys and sensor data, the Investigators aim to identify novel types of clinical data that can be used as digital biomarkers with complementary clinical value as compared to the traditional diagnostic methods and techniques.

In this feasibility study a number of digital biomarkers will be applied to test their technical reproducibility/stability and meaningfulness to patients.

DETAILED DESCRIPTION:
Multiple Sclerosis (MS) is a chronic inflammatory disease of the central nervous system (CNS) causing focal lesions of demyelination and diffuse neurodegeneration in the grey and white matter of the brain and spinal cord, leading to physical and cognitive disability. Currently there is a limited number of relevant biomarkers available in patients with MS, such as clinical, imaging or biological measures. Patient history and neurologic examination in combination with magnetic resonance imaging (MRI), evoked potentials and analysis of serum and cerebrospinal fluid (CSF) are the gold standard of diagnosis and mainly patient history, neurologic examination and MRI are used for patient monitoring. However, their prognostic value on a patient level is still very limited. Therefore, the scientific community and patients are in need for new and more reliable biomarkers, especially biomarkers of disease progression in order to adapt therapeutic approaches on an individual level. Digital biomarkers have the potential to fill this gap allowing for quasi-continuous measures that might be more informative than episodically collected conventional data concerning the impact of the disease on activities of daily living.

The Investigators have developed the dreaMS App, a data communication platform collecting data from the patients' mobile devices (smartphone and wearables). Through the use of app-based tests, surveys and sensor data, the Investigators aim to identify novel types of clinical data that can be used as digital biomarkers with complementary clinical value as compared to the traditional diagnostic methods and techniques.

In this feasibility study a number of digital biomarkers will be applied to test their technical reproducibility/stability and meaningfulness to patients and to select the most informative for the planned validation study.

ELIGIBILITY:
Patients with MS

Inclusion Criteria:

* Age 18-70
* Diagnosed with MS according to the revised McDonald criteria 2017, all clinical forms inclusive (CIS, RRMS, SPMS, PPMS)
* EDSS ≤ 6.5
* In possession of a smart phone

Exclusion Criteria:

* Age <18 and > 70
* EDSS > 6.5
* Other clinically significant concomitant disease states (e.g., renal failure, severe hepatic dysfunction, severe/unstable cardiovascular disease, progressive cancer, etc.)
* Known or suspected non-compliance, drug or alcohol abuse
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc.
* Women who are pregnant or breast feeding
* Not in possession of a smart phone

Healthy Volunteers

Inclusion Criteria:

* Age 18-70
* In possession of a smart phone

Exclusion Criteria:

* Age <18 and > 70
* Diagnosis of MS
* Clinically significant concomitant disease states (e.g., renal failure, severe hepatic dysfunction, severe/unstable cardiovascular disease, progressive cancer, etc.)
* Known or suspected non-compliance, drug or alcohol abuse
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc.
* Women who are pregnant or breast feeding
* Not in possession of a smart phone

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2020-10-05 (Actual); Primary Completion 2021-02-26 (Actual); Study Completion 2021-02-26 (Actual)

PRIMARY OUTCOMES:
Test Reliability of digital biomarkers measured by Intra Class Correlation | 6 weeks
  Number of digital biomarkers tested with an Intra Class Correlation of at least 0.6 if repeated 10 times
Test Reliability of digital biomarkers measured by Coefficient of variation | 6 weeks
  Number of digital biomarkers tested with a coefficient of Variation of less than 20% if repeated 10 times
Determination of user acceptance of each digital biomarker with regards to acceptance based on a questionnaire using a likert scale | 6 weeks
  Number of digital biomarkers tested with a good acceptance reflected by a mean response of more than 3 on a likert scale.

CONTACTS AND LOCATIONS:
Overall Officials: Ludwig Kappos, MD, Principal Investigator — University Hospital Basel and RC2NB
Locations (1):
- RC2NB, Basel, Switzerland

REFERENCES:
- [Derived] Pless S, Woelfle T, Naegelin Y, Lorscheider J, Wiencierz A, Reyes O, Calabrese P, Kappos L. Assessment of cognitive performance in multiple sclerosis using smartphone-based training games: a feasibility study. J Neurol. 2023 Jul;270(7):3451-3463. doi: 10.1007/s00415-023-11671-9. Epub 2023 Mar 23. PMID 36952010
- [Derived] Woelfle T, Pless S, Reyes O, Wiencierz A, Feinstein A, Calabrese P, Gugleta K, Kappos L, Lorscheider J, Naegelin Y. Reliability and acceptance of dreaMS, a software application for people with multiple sclerosis: a feasibility study. J Neurol. 2023 Jan;270(1):262-271. doi: 10.1007/s00415-022-11306-5. Epub 2022 Aug 30. PMID 36042020